CLINICAL TRIAL: NCT05614037
Title: Felodipine Controlled Release Tablets and Felodipine Sustained Release Tablets in Healthy Subjects Under Fasting State: Single Dose, Randomized, Open, 2-treatment，2-period，Crossover Comparative Pharmacokinetic Study
Brief Title: Felodipine Controlled Release Tablets and Felodipine Sustained Release Tablets in Healthy Subjects Under Fasting State Comparative Pharmacokinetic Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Overseas Pharmaceuticals, Ltd. (Industry)
Collaborators: Guangzhou Kangqi Medical Technology Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: YYKQ-202207
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-10

CONDITIONS: Hypertension
Keywords: Felodipine; Hypertension; Healthy Volunteers; morning surge
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Test preparation (T) : Felodipine Controlled Release Tablets Specification: 5 mg Batch number: 22090301 Content: 100.8% Valid until: September 2024 Storage conditions: sealed, room temperature (10~30℃) Manufacturer: Overseas Pharmaceuticals, Ltd. Supplier: Overseas Pharmaceuticals, Ltd. Reference preparation (R) :Felodipine Modified-release tablets(trade name: plendil ®) Specification: 5 mg Batch number: 2204 a11 Content: 99.1% Valid until March 2025 Storage conditions: below 25℃ Manufacturer: AstraZeneca AB Supplier: Overseas Pharmaceuticals, Ltd.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Felodipine Controlled Release Tablets (Experimental): Test preparation (T) :Felodipine Controlled Release Tablets Specification: 5 mg Batch number: 22090301 Content: 100.8% Valid until: September 2024 Storage conditions: sealed, room temperature (10~30℃) Manufacturer: Overseas Pharmaceuticals, Ltd. Supplier: Overseas Pharmaceuticals, Ltd. Usage: Oral, 1 tablet at a time, once a day. Take it before bed and swallow it with water. Do not break, press or chew the pill.
  Interventions: Drug: Felodipine sustained release tablets (trade name: plendil®)
- Felodipine Modified-release Tablets (trade name:plendil ®) (Active Comparator): Reference preparation (R) : Felodipine Modified-release Tablets (trade name:plendil ®) Specification: 5 mg Batch number: 2204 a11 Content: 99.1% Valid until March 2025 Storage conditions: below 25℃ Manufacturer:AstraZeneca AB Supplier: Overseas Pharmaceuticals, Ltd. Usage: Oral, 1 tablet at a time, once a day. Take it before bed and swallow it with water. Do not break, press or chew the pill.
  Interventions: Drug: Felodipine Controlled Release Tablets

INTERVENTIONS:
Drug: Felodipine sustained release tablets (trade name: plendil®) — Reference preparation (R) : Felodipine sustained release tablets (trade name: plendil ®) Specification: 5 mg Batch number: 2204 a11 Content: 99.1% Valid until March 2025 Storage conditions: below 25℃ Manufacturer: AstraZeneca AB Supplier: Overseas Pharmaceuticals, Ltd. Usage: Oral, 1 tablet at a time, once a day. Take it before bed and swallow it with water. Do not break, press or chew the pill.
  Arms: Felodipine Controlled Release Tablets
Drug: Felodipine Controlled Release Tablets — Test preparation (T) :Felodipine Controlled Release Tablets Specification: 5 mg Batch number: 22090301 Content: 100.8% Valid until: September 2024 Storage conditions: sealed, room temperature (10~30℃) Manufacturer: Overseas Pharmaceuticals, Ltd. Supplier: Overseas Pharmaceuticals, Ltd. Usage: Oral, 1 tablet at a time, once a day. Take it before bed and swallow it with water. Do not break, press or chew the pill.
  Arms: Felodipine Modified-release Tablets (trade name:plendil ®)

SUMMARY:
Felodipine Controlled Release Tablets and Felodipine Modified-release Tablets in Healthy Subjects Under Fasting State: Single Dose, Randomized, Open, 2-treatment，2-period，Crossover Comparative Pharmacokinetic Study

Main research objectives:

Felodipine Controlled Release Tablets(strength: 5 mg) developed by Overseas Pharmaceuticals, Ltd., and Felodipine Modified-release Tablets (strength: 5 mg) produced by AstraZeneca AB., trade name: The pharmacokinetic parameters of the test preparation and the reference preparation in healthy subjects under fasting state were investigated and compared.

Secondary research objectives:

To observe the safety of test preparation and reference preparation in healthy subjects.

DETAILED DESCRIPTION:
The subjects were randomly assigned in a 1:1 ratio to one of two sequential administration groups (group T-R, group R-T). In the first cycle, 8 subjects took the test formulation (T) 5 mg/tablet by fasting, and the other 8 subjects took the reference formulation (R) 5 mg/tablet by fasting, with about 240 mL warm water. The drug was crossed over after 14 days. Phase I trial site pharmacists assigned study drugs to each phase according to the randomization list.

Sixteen healthy subjects were randomly divided into two groups, T-R group and R-T group, with 8 cases in each group. The enrolled subjects entered the phase I observation room one day before the administration of each cycle, and were required to fast for more than 10 hours from the day before to the morning of the administration. After a blank blood sample was collected on the morning of administration, the study drug was administered in the fasting state. The standard meal was taken 4 hours after administration. Each week was performed at 0 h before administration (within 1.5 h before administration) and 0.5 h, 1.0 h, 1.5 h, 2.0 h, 2.5 h, 3.0 h, 3.5 h, 4.0 h, 4.5 h, 5.0 h, 5.5 h, 6.0 h, 6.5 h, 7.0 h, 7.5 h, 8.0 h, 8.5 h, 9.0 h, 10.0 h, 12.0 h, 24.0 h, 48.0 h, 72.0 h, a total of 24 blood sampling points were collected from the upper limb vein.

Vital signs (including body temperature (frontal temperature), pulse and blood pressure) were measured at 0 h before administration (within 1.5 h before administration) and 4.0± 0.5 h, 8.0± 0.5 h, 24.0± 1.0 h, 48.0± 1.0 h and 72.0± 1.0 h after administration. The operation procedure of the second cycle is the same as that of the first cycle. In the second cycle, the subjects were required to take physical examination, vital signs examination, electrocardiogram and laboratory examination on the day after the end of sampling.

If a subject has an AE during the trial, the investigator should try to follow the subject until the adverse event resolves, or returns to the screening level, or the subject's condition is stable.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is fully aware of the purpose, nature, method and possible adverse reactions of the study, voluntarily acts as a subject, and signs informed consent prior to the commencement of any study procedure.
2. Healthy subjects (male or female) aged 18 years or older.
3. Male weight ≥50.0 kg, female weight ≥45.0 kg; Body mass index (BMI) was in the range of 19.0 to 26.0 kg/m2 (including the critical value).
4. From the signing of informed consent to 6 months after the end of the study, they had no fertility plan, voluntarily took appropriate and effective contraceptive measures, and had no sperm and egg donation plan.
5. The subjects were able to communicate well with the researchers and understood and complied with the requirements of the study.

Exclusion Criteria:

1. Allergic disposition or a history of food or drug allergy or other allergic diseases (asthma, urticaria, eczema dermatitis, etc.) that researchers deem clinically significant; Or allergic to any component of felodipine.
2. Patients with poor vascular puncture conditions, or who cannot tolerate venipunction, or who have a history of fainting needles and fainting blood.
3. Patients with gingivitis and periodontitis.
4. Previous history of compensatory heart failure, acute myocardial infarction, unstable angina pectoris.
5. lactose intolerance, or galactose intolerance, lactase deficiency, glucose-galactose malabsorption.
6. Patients with confirmed hypotension or history of postural hypotension.
7. The presence of cardiovascular, blood, liver, kidney, endocrine, respiratory, digestive, nervous, psychiatric, immune, skin, metabolic disorders and other systemic diseases considered clinically significant by researchers, or a chronic or severe history of these diseases; Or a history of surgery that may affect drug absorption and metabolism.
8. Physical examination, vital signs examination, 12-lead electrocardiogram and laboratory examination were abnormal and clinically significant as judged by the study physician.
9. Positive for human immunodeficiency virus (HIV) antibody, hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or treponema pallidum antibody (Anti-TP).
10. Pregnant women, breastfeeding women, or women of childbearing age who have unprotected sex or pregnancy test positive within 14 days before the planned dose.
11. Those who received vaccines (other than COVID-19 vaccine) within 3 months prior to screening, or who received COVID-19 vaccine within 1 week prior to screening, or who plan to receive any vaccines during the trial or within 1 week after the study ends;
12. Those who have donated blood/lost blood ≥400 mL in the 3 months prior to screening or who have received blood transfusions or used blood products, or who intend to donate blood (including blood components) during or 3 months after the end of the trial.

    Previous drug use:
13. Those with a history of drug abuse or who have tested positive for drugs and used drugs in the six months prior to screening, including methylenedioxymethamphetamine (ecstasy), methamphetamine (meth), ketamine, morphine, and THC (marijuana).
14. Drugs that inhibit or induce liver metabolism of drugs (such as inducers: barbiturates, carbamazepine, phenytoin, rifampicin, St. John's wort, etc.) were used within 28 days before the initial administration; Inhibitors: cimetidine, cyclosporine, pyrrole antifungal drugs (itraconazole, ketoconazole), macrolides antibiotics (erythromycin), HIV protease inhibitors, etc.); Or any other medication including prescription drugs, over-the-counter drugs, functional vitamins, health products, or Chinese herbs used in the 14 days prior to administration.

    Diet and smoking and alcohol consumption:
15. People who have difficulty swallowing or have special requirements for diet and cannot accept unified diet.
16. Habitual long-term consumption of excessive (more than 8 cups a day, 1 cup =250 mL) of food or drink containing caffeine (such as coffee, strong tea, cola, chocolate, etc.), or ingestion of food or drink containing caffeine within 72 hours before the first medication, or can not be interrupted during the trial.
17. People who consumed purine-rich foods (such as anchovies, sardines, beef liver, beef kidney, etc.) or products containing grapefruit, grapefruit juice, grape juice, menthol within 48 hours before administration, or planned intake or could not be interrupted during the trial.
18. Those who had started a significantly abnormal diet (e.g., diet, low sodium) within 4 weeks prior to screening.
19. Excessive smoking within 6 months prior to screening (mean ≥5 doses/day) or within 48 hours prior to the first dose, or unable to stop using any tobacco products during the trial.
20. those who have a history of alcoholism or are regular drinkers in the six months prior to screening, that is, drinking more than 14 units of alcohol per week (1 unit =360 mL beer with 5% alcohol by volume or 45 mL spirits with 40% alcohol by volume or 150 mL wine with 12% alcohol by volume), Or consumed alcohol or food or beverages within 48 hours before the first dose, or tested positive for alcohol on the day of the first cycle check-in, or were unable to stop alcohol consumption during the study period.

    Other:
21. Participants who had participated or were participating in clinical trials of other drugs (defined as having used investigational drugs) in the 3 months prior to screening.
22. Subjects who were assessed by the investigator for other factors unsuitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from time zero to the time of the last quantifiable plasma concentration of the period (AUC0-last) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation) of AUC0-last within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Area under the curve from time zero to infinity (AUC0-inf) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of AUC0-inf within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Peak concentration at each treatment period (Cmax,tp) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of Cmax,tp within [0.8, 1.25] range will be used to determine the result of bioequivalence.

SECONDARY OUTCOMES:
Peak concentration of the first dosing (Cmax) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Time to reach peak concentration of the first dosing (Tmax) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Terminal half-life (T1/2) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Mean residence time (MRT) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Centre of Dongguan Kanghua Hospital, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No